CLINICAL TRIAL: NCT04724525
Title: The Effect of Changes in Power and Cylinder Axis on Vision Quality, Satisfaction and Vision Acceptability of People With Mild-Medium Astigmatism With Toric Soft Contact Lenses (LKL)
Brief Title: Changes in Power and Cylinder Axis of Toric Soft Contact Lenses (LKL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dwie Aprina, Principal investigator, Indonesia University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 20-070-0813
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Visual Acuity Reduced Transiently
Keywords: Toric soft contact lens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: soft contact lens Toric — soft contact lens toric with different axis and power that use in human's eye

SUMMARY:
Astigmatism is a common refractive error resulting from a toric-surfaced cornea which using a toric soft contact lens could be one of the therapy options. Due to the numerous possible combinations between sphere powers, cylinder powers, and cylinder axes, manufacturers of disposable soft toric contact lenses limit their toric lens range, while still aiming to cater to the majority of astigmatic patients. Due to that reason, the possibility of astigmatism patients getting a different combination of power and axis with toric soft contact lenses sold on the market will be high due to SKU limitations. This research aims to ascertain the impact of altering cylinder power and axis on visual quality and convenience in astigmatism participants using toric soft contact lens. The study was conducted at Kirana Ciptomangunkusumo Hospital, Jakarta, starting in April 2020. The study is a prospective, randomized, participant-masked, crossover clinical trial where the participants were tested for the following conditions on different days using full spherocylinder correction and under-correction by 0.25, 0.50, and 0.75 DC while maintaining spherical equivalence. Axis was also misaligned between -30° and +30°, in 10° steps. For each visit, the patient was examined visual acuity, contrast visual acuity using the Pelli-Robson, and assessed patient comfort using the VAS method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 - 35 years
2. Patients who do not have a spherical size (plano) to mild-moderate myopia (-1.00 D to -6.00 D) with age over 18 years
3. Minimum astigmatism component ≥0.75 D and maximum ≤ 3 D in one eye
4. The best visual acuity after corrected by LKL Torik is better or equal to 6/15

Exclusion Criteria:

1. History of previous intraocular surgery.
2. History of contact lens use in the last 6 months.
3. history of dry eyes, uveitis, glaucoma and corneal and conjunctival disorders
4. posterior segment abnormalities that reduce the quality of vision
5. Patients with contraindications to wearing contact lenses
6. There are no toric LKLs with exactly the strength and axes required by the patient

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Visual Acuity | when using a contact lens (0 day,7 days, 14 days)
  Visual acuity was measured using a Snellen chart at a distance of 6 meters by the researcher (DA) at Refractive Poly

SECONDARY OUTCOMES:
Change in Contrast sensitivity | when using a contact lens (0 day,7 days, 14 days)
  Value obtained on examination of the Pelli Robson Chart in Poly Neurooftlamology. Examination conducted by researchers (DA).
Visual Clarity | when using a contact lens (0 day,7 days, 14 days)
  Values were obtained by the VAS method. Research subjects were asked to name a number from 1-10 (score 1 indicates poor clarity, 10 indicates good clarity) to assess visual clarity
Visual Satisfaction | when using a contact lens (0 day,7 days, 14 days)
  Values were obtained by the VAS method. The research subjects were asked to name a number from 1-10 (a score of 1 indicates dissatisfaction, 10 indicates very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia